CLINICAL TRIAL: NCT05924958
Title: College of Pharmacy, Xinjiang Medical University
Brief Title: Clinical Study on the Immunomodulatory Effect of Eprolidone on Patients With Chronic Heart Failure
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cheng LuFeng,Principal Investigator (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Sponsor-Investigator, Cheng LuFeng,Principal Investigator, College of Pharmacy, Xinjiang Medical University, Xinjiang Medical University
Organization: Xinjiang Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LFCheng
Record Dates: First submitted 2023-06-06; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Chronic Heart Failure Patients

STUDY DESIGN:
Intervention Model Description: Conventional treatment group Eprolidone group
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eprolidone intervention in patients with chronic heart failure (Experimental): The Pulidone group received conventional medication combined with 25 mg/day of Eprolidone, gradually increasing to 50 mg/day for 4 consecutive weeks
  Interventions: Drug: Eprolidone
- Patients in the conventional treatment group (No Intervention): Other conventional anti chronic heart failure drugs for the conventional treatment group taking non aldosterone receptor blockers

INTERVENTIONS:
Drug: Eprolidone — This study assessed the effect of eplerenone on circulating Treg cells in patients with chronic heart failure by detecting the level of aldosterone in venous blood and the activity of Treg cells and the level of inflammatory factors related to it after taking drugs.
  Arms: Eprolidone intervention in patients with chronic heart failure

SUMMARY:
Chronic heart failure has a high incidence, mortality rate, and disability rate. There are approximately 4 million heart failure patients among adults aged 35-74 in China, which has become a major public health issue. In this context, accelerating the development of drugs for treating chronic heart failure has become an urgent and urgent problem to be solved. Therefore, revealing the pathogenic mechanism of chronic heart failure, finding specific drug intervention targets, conducting personalized and precise diagnosis and treatment, reducing the economic burden of patients, and promoting national economic development have significant practical significance and far-reaching strategic impact. Heart failure, as the final stage of various cardiovascular diseases, is difficult to recover once it occurs, so it is of great benefit to achieve "early detection and treatment" for heart failure. At present, biomarkers are mainly used for the diagnosis and prognosis of heart failure, and there are very few biomarkers that provide early warning information. Therefore, it is urgent to find biomarkers that can provide early warning effects. This project focuses on the effect of Eprolidone on the activity of regulatory T cells (Treg), expanding the selection of heart failure treatment drugs, improving drug efficacy, avoiding ineffective treatment, and reducing adverse reactions of the drugs. By carrying out high-quality and precise treatment, we aim to promote the update of the diagnosis and treatment guidelines for chronic heart failure, and provide treatment plans for the prevention and treatment of chronic heart failure and the formulation and adjustment of national medical and health policies.

DETAILED DESCRIPTION:
Recruit participants subjects and sign a written informed consent form. Randomly divide the participants into a conventional treatment group and an epridone group. The conventional treatment group received other conventional anti chronic heart failure drugs that were not aldosterone receptor blockers, and the baseline was taken. The epridone group received conventional medication combined with 25 mg/day of epridone, gradually increasing to 50 mg/day for 4 consecutive weeks.The participants' venous blood was drawn once a week to test the participants' cardiac function and related immunological indicators.Regularly follow up participants to compare adverse reactions and clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form, NYHA Level I, Level II Ш The left ventricular ejection fraction (LVEF) measured by radionuclide ventriculography (RNVG) after diagnosis of chronic congestive heart failure (CHF) is ≤ 45%.

Exclusion Criteria:

* Age<18 or>80, serum creatinine level>2.5 mg/deciliter, blood potassium level>5.0 mmol/liter, surgical treatment for valvular heart disease, contraindications to the study drug, use of other aldosterone receptor antagonists, malignant tumors and other life-threatening non cardiac diseases, legally incapacitated patients, history of drug and alcohol abuse, pregnant and postpartum women, and women breastfeeding during the study period. The subjects were divided into a conventional treatment group and an epridone group, with the conventional treatment group taking other conventional anti chronic heart failure drugs other than aldosterone receptor blockers as the baseline. The epridone group received conventional medication combined with 25 mg/day of epridone, gradually increasing to 50 mg/day for 4 consecutive weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Expression of Kv1.3 channel protein in Treg cells in circulating blood | 4 weeks
  Detection of Treg cell activity in venous blood of patients
Levels of aldosterone in blood circulation （pg/mL) | 4 weeks
  Detection of aldosterone in venous blood of patients by ELISA
The levels of IL-10 and TGF-β in blood circulation （pg/mL) | 4 weeks
  Detection of plasma inflammatory factors in subjects

SECONDARY OUTCOMES:
Detection of left ventricular Ejection fraction by echocardiography | 4 weeks
  Echocardiographic detection of cardiac function in patients